CLINICAL TRIAL: NCT02773966
Title: Intraoperative Radiotherapy During Kyphoplasty/Vertebroplasty (Kypho-IORT) Versus EBRT in the Treatment of Painful Vertebral Metastases - a Randomized Prospective Phase III Study -
Brief Title: Kypho-IORT vs. EBRT in Spinal Metastases
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Frederik Wenz, Prof. Dr. Frederik Wenz, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kypho-IORT/EBRT
Record Dates: First submitted 2016-05-04; First posted 2016-05-16 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Metastasis
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Kypho-IORT (Experimental): balloon kyphoplasty/vertebroplasty + intraoperative radiotherapy
  Interventions: Radiation: Kypho-IORT
- Arm B: EBRT (Active Comparator): external beam radiotherapy with 30 Gy during 10 days (3 Gy/day)
  Interventions: Radiation: EBRT

INTERVENTIONS:
Radiation: Kypho-IORT — During kyphoplasty/vertebroplasty a intraoperative radiotherapy of the affected vertebrae is done with a miniature X-ray generator (INTRABEAM®, Carl Zeiss, Surgical, Oberkochen, Germany). The prescription dose will be 8 Gy in a distance of 13 mm from the isocenter of the radiation source. IORT will take about five minutes. After radiation the applicator will be removed and the operation will be finished as usual.
  Arms: Arm A: Kypho-IORT
Radiation: EBRT — The external beam radiotherapy will be usually carried out as an outpatient procedure. All patients will receive a planning CT before the first irradiation. EBRT will be performed with 30 Gy, added in 3 Gy per fraction or 8 Gy single dose (only for international study centers, not permitted in Germany) on a conventional linear accelerator (LINAC).
  Arms: Arm B: EBRT

SUMMARY:
The objective of this randomized phase III study is to test the superiority of Kypho-IORT compared to EBRT with regard of time to pain reduction in patients with painful vertebral metastases. Therefore patients will receive intraoperative radiotherapy (8 Gy with Intrabeam System/Carl Zeiss) during kyphoplasty (Arm A) or external beam radiotherapy with 30 Gy, added in 3 Gy per fraction on a conventional linear accelerator or 8 Gy single dose (only for international study centers, not permitted in Germany) (Arm B).

DETAILED DESCRIPTION:
Due to optimized therapies life expectancy of patients with metastasizing cancer increases. Bone metastases affect 10% - 30% of all cancer patients, especially located in the vertebral column. The main clinical problems are back pain and an increased risk of pathological fracture. Therefore optimized palliative treatments to improve quality of life are necessary.

External beam radiotherapy (EBRT) is a well-established treatment option for patients with spinal metastases. EBRT often results in an adequate pain relief with good local tumor control . Of the retrospective series that described pain outcome mentioned in the systematic review by Gerszten et al., a mean of 70% of patients had improvement in pain after radiation therapy. The mean rate of local control was 77%. Although EBRT is the standard treatment for painful vertebral metastases, the optimal dose fraction schedule or the optimal standard dose has not been established. Different fractionation schedules of EBRT are discussed in a recently published review. Literature data confirm time to pain reduction of about 8-10 days after EBRT.

Balloon kyphoplasty is another valuable treatment option for patients with painful and instable metastases to the vertebral column. In the recent published trial by Berenson et al. 134 patients with vertebral compression fractures were enrolled and randomly assigned to kyphoplasty or non-surgical management. The study found that patients treated with kyphoplasty had a significant reduction of back pain after seven days. Nevertheless kyphoplasty has no direct anticancer effect and external beam radiotherapy has to follow to avoid early regrowth. But EBRT after kyphoplasty or EBRT alone takes up to 2-4 weeks. This long treatment period can often be a mental and physical strain. Moreover patients with simultaneous visceral metastases often need chemotherapy which cannot be applied concurrently to radiotherapy due to the risk of potentiated toxicity. To reduce treatment time and increase quality of life novel techniques like kyphoplasty combined with other physical methods are under development. Recently published trials showed good results relating to pain relief and local tumor control in patients with spinal metastases treated with kyphoplasty combined with intravertebral administration of 153Samarium or interstitial implantation of 125I seeds. Therefore we developed a novel approach to deliver intraoperative radiotherapy during kyphoplasty (Kypho-IORT). Based on our recently published reports Kypho-IORT is a technical feasible new treatment option without severe side effects. We observed an excellent pain relief. At the first postoperative day improvement of pain was observed in 11 of 16 (69%) patients and no change in 5 of 16 (31%) patients. During further follow-up, improvement of pain was seen in 75% - 83% of the patients compared to the preoperative status. According to these results a dose escalation study has been initiated, which has been completed (NCT 01280032). According to the results of this study a dose of 8 Gy in 10 mm depth from the applicator surface (correlates to a dose prescription from the isocenter of the radiation source of 8 Gy in 13 mm) is recommended for further Kypho-IORTs.

According to this the aim of this planned phase III study is to test the superiority of kyphoplasty or vertebroplasty + IORT (in the following abbreviated as Kypho-IORT) compared to EBRT with regard to time to pain reduction at defined points in time (day 1, week 2, 6 weeks after start of treatment).

We assume a pain reduction of VAS-3 points at day one (first day after Kypho-IORT, one day after the first EBRT) for 40% of the patients after Kypho-IORT vs. 5% of the patients after EBRT under standard pain medication (no change of the pretherapeutic pain medication 12 h after Kypho-IORT or rather 24 h after the first EBRT). Each study arm needs 22 patients, to reach an alpha of 0, 05 and a power of 0,817. Plus a dropout rate of 20% at least 54 patients have to be recruited.

All patients with spinal metastases who present for treatment will be given, if these have not been done in advance: a MRI and a CT of the total spine and a clinical examination, especially a neurological examination.

Kypho-IORT will be carried out under general anaesthesia like the standard procedure with minor modifications. All patients will be placed in prone position on a radiolucent table. For intraoperative radiotherapy (IORT) the Intrabeam System (Carl Zeiss Surgical, Oberkochen, Germany) will be used. In order to carry out the intraoperative radiation therapy, working cannulas are inserted into the affected vertebral body in a normal bipedicular procedure, special sleeves are inserted monopedicularly. These serve as guides for the radiation applicator. After checking the correct positioning of the working cannulas using fluoroscopic guidance, the specially designed applicator is placed precisely in the vertebral body. Documentation of the location of the tip of the INTRABEAM System should be performed whenever possible using bi-planar X-rays.

After verification the selected dose of 8 Gy in a depth of 13 mm from the isocenter of the radiation source is applied for a period of approximately 5 minutes.

After completion of the radiation therapy, the radiation unit including the applicator is removed and the operation is concluded in accordance with standard procedure.

The external beam radiotherapy will be usually carried out as an outpatient procedure. All patients will receive a planning CT before the first irradiation. EBRT will be performed with 30 Gy, added in 3 Gy per fraction or 8 Gy single dose (only for international study centers, not permitted in Germany) on a conventional linear accelerator (LINAC). During EBRT, patients are routinely seen once weekly by physicians and evaluated for adverse reactions.

Before treatment the registration form has to be filled out including the following items:

* evaluation of inclusion and exclusion criteria,
* anamnesis (size, weight, Karnofsky Index, standard pain medication, concomitant illnesses),
* objectification of the patient's current pain situation using the Visual Analog Scale (VAS) local and in general,
* primary tumor,
* localization and size of the vertebral body metastases
* quality of life assessment (EORTC QLQ-C30, EORTC QLQ-BM22). Moreover all patients receive an MRI and a CT of the spine and a neurological examination.

Follow-up visits will be scheduled after 6 weeks, then after 3 months, then every 6 months up to 5 years. At each follow-up the following information will be documented:

* weight,
* Karnofsky Index,
* general progress/regress of underlying illness,
* standard pain medication
* pain level based on the VAS (in general, local).

Furthermore, an inspection of the surgical scar to exclude wound healing problems and a neurological examination to document any functional impairment due to spinal cord or nerve damage will be carried out. To assess skin toxicity, photographic documentation of the surgical scar/irradiation field will be carried out. For documentation of osteoradionecrosis, pathological fractures and relapses a MRI or CT examinations will be carried out. The evaluation of the MRI or CT examinations will be performed by the radiologists of the respective participating clinic, or in the case of externally prepared images, by the radiologists of the medical practice. To document Quality of Life, the patients will be requested to complete two questionnaires of the European Organization for Research and Treatment of Cancer (EORTC QLQ-C30, EORTC QLQ-BM22) before Kypho-IORT/EBRT and during the follow-up examinations. Answering the questions will take approximately 10 minutes. The follow-up and documentation of patient specific data will end 5 years after therapy.

Classification and graduating of side effects are rated by "Common Toxicity Criteria" (CTCv4.0) of the National Cancer Institute. To document acute toxicities after Kypho-IORT, a physical examination including in particular an inspection of the surgical scar and an evaluation of the current pain level (VAS) will be performed one day and 2 weeks after Kypho-IORT. Moreover a conventional X-ray of the affected section of the spine will be performed one day after Kypho-IORT. One day after the first EBRT and after the last EBRT, same-day, a physical examination and an evaluation of the current pain level (VAS) will be performed to document acute toxicities. Moreover during EBRT, patients are routinely seen once weekly by physicians and evaluated for adverse reactions. If necessary, any occurring acute reactions will be documented upon discharge from the hospital and checked at the follow-up appointments.

The acquisition of late toxicities will be done based on the LENT SOMA score. To document the late toxicities, follow-up examinations with magnetic resonance imaging or computer tomography, as well as another physical examination will be performed. Moreover a photographic documentation of the surgical scar/irradiation field will be carried out to assess skin toxicity.

Serious adverse events (SAEs) are defined as any event that is fatal, life threatening, causes or prolongs hospitalization; causes disability or incapacity or requires medical intervention to prevent permanent impairment or damage, or any grade 4 toxicity. Only radiation or surgery related SAEs should be reported. Hospitalization for performing protocol-required procedures is not classified as an SAE. Hospitalization for disease-related procedures (surgery, imaging, laboratory tests) or any procedures planned before entry into the study are not considered SAEs. Hospitalizations for social reasons in the absence of an adverse event are not classified as SAEs either. Furthermore radiation or surgery related SAEs requiring therapy should be documented (e.g. antibiotics, re-surgery).

In case of death an autopsy should be done to clarify the cause of death. The trial will be carried out in compliance with the protocol, the principles laid down in the declaration of Helsinki, version as of October 1996 (as long as local laws do not require to follow other versions), in accordance with the ICH Harmonised Tripartite Guideline for Good Clinical Practice (GCP), the harmonized standards for Medical Devices (ISO 14155) and all other applicable regulatory requirements (local, regional and global). Standard medical care (prophylactic, diagnostic and therapeutic procedures) remains in the responsibility of the treating physician of the patient.

This study is approved by the local ethics committee and the Federal Office of Radiation Protection.

The informed consent is performed written and verbally by the responsible physician. The informed consent is done at least 24 h before treatment. During the education the physician has to indicate that a withdrawal is possible at each time and does not result in disadvantages for the patient.

Treatment of the patient must be discontinued if one or more of the following criteria apply:

* revocation of the patient's declaration of informed consent
* lack of compliance
* discontinuation of the therapy for other reasons deemed necessary by the responsible physician (unfavorable intraoperative geometry)
* Grade IV skin toxicity, i.e. skin necroses that require surgical intervention
* Grade IV bone toxicity, i.e. aseptic bone necroses that require surgical intervention
* Grade IV nervous system toxicity, i.e. paresis When therapy is discontinued, the reasons for discontinuing patient participation in the study must be listed in the patient's file.

The steering committee is allowed to close the study ahead of schedule.

Other termination criteria include:

* insufficient patient recruitment
* unexpectedly severe toxicities (second Grade IV toxicity within the study)
* unexpected findings which prevent the continuation of the study for ethical and/or medical reasons (new benefit/risk analysis)

ELIGIBILITY:
Inclusion Criteria:

* ≥ 50 years
* Karnofsky Index ≥ 60
* Initial pain score using the VAS ≥ 3 under standard pain medication
* Histological or by imaging proven painful osteolytic metastases (max. 4 treatable vertebrae) of the thoracic/lumbar spine, which are accessible for Kypho-IORT
* Written informed consent obtained
* Exclusion Criteria:
* Previous local treatment (irradiation, surgery)
* Cranial site of the metastasis above T4
* Pathological fracture with sintering >50%
* Purely osteoblastic metastasis
* Intraspinal extension
* Erosion of the bony borders of the vertebra which make a cement filling difficult, rated by the treating surgeon
* Tumor expansion to dorsal vertebral structures (pedicle, lamina)
* Pregnancy/lactation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-11-12 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
pain evaluation | day 1
  Evaluation of the percentage of patients with a pain reduction of VAS-3 points after Kypho-IORT vs. EBRT at day 1 (one day after Kypho-IORT; one day after the first EBRT)

SECONDARY OUTCOMES:
pain evaluation | week 2, 6 weeks after start of treatment
  Evaluation of the percentage of patients with a pain reduction of VAS-3 at week 2 and 6 weeks after start of treatment
local recurrence rate | 6 weeks, then after 3 months, then every 6 months up to 5 years
  local recurrence diagnosed by a MRI or CT scan
Quality of life (QoL) questionaire | before start of therapy and then 6 weeks, then after 3 months, then every 6 months up to 5 years
  Assessed by European Organization for Research and Treatment (EORTC)-Quality of Life questionaires (QLQ-C30/BM22)
Overall survival | 12 Months
  Overall survival will be calculated from the date of Kypho-IORT/start of EBRT until the date of death from any cause or date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Giordano, MD, Principal Investigator — Universitätsmedizin Mannheim
Locations (1):
- Department of Radiotherapy University Hospital Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerszten PC, Mendel E, Yamada Y. Radiotherapy and radiosurgery for metastatic spine disease: what are the options, indications, and outcomes? Spine (Phila Pa 1976). 2009 Oct 15;34(22 Suppl):S78-92. doi: 10.1097/BRS.0b013e3181b8b6f5. PMID 19829280
- [Background] Souchon R, Wenz F, Sedlmayer F, Budach W, Dunst J, Feyer P, Haase W, Harms W, Sautter-Bihl ML, Sauer R; German Society of Radiation Oncology (DEGRO). DEGRO practice guidelines for palliative radiotherapy of metastatic breast cancer: bone metastases and metastatic spinal cord compression (MSCC). Strahlenther Onkol. 2009 Jul;185(7):417-24. doi: 10.1007/s00066-009-2044-2. Epub 2009 Aug 28. PMID 19714302
- [Background] Berenson J, Pflugmacher R, Jarzem P, Zonder J, Schechtman K, Tillman JB, Bastian L, Ashraf T, Vrionis F; Cancer Patient Fracture Evaluation (CAFE) Investigators. Balloon kyphoplasty versus non-surgical fracture management for treatment of painful vertebral body compression fractures in patients with cancer: a multicentre, randomised controlled trial. Lancet Oncol. 2011 Mar;12(3):225-35. doi: 10.1016/S1470-2045(11)70008-0. Epub 2011 Feb 16. PMID 21333599
- [Background] Schneider F, Greineck F, Clausen S, Mai S, Obertacke U, Reis T, Wenz F. Development of a novel method for intraoperative radiotherapy during kyphoplasty for spinal metastases (Kypho-IORT). Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):1114-9. doi: 10.1016/j.ijrobp.2010.07.1985. Epub 2010 Oct 8. PMID 20934272
- [Background] Wenz F, Schneider F, Neumaier C, Kraus-Tiefenbacher U, Reis T, Schmidt R, Obertacke U. Kypho-IORT--a novel approach of intraoperative radiotherapy during kyphoplasty for vertebral metastases. Radiat Oncol. 2010 Feb 11;5:11. doi: 10.1186/1748-717X-5-11. PMID 20149237
- [Background] Schmidt R, Wenz F, Reis T, Janik K, Bludau F, Obertacke U. Kyphoplasty and intra-operative radiotheray, combination of kyphoplasty and intra-operative radiation for spinal metastases: technical feasibility of a novel approach. Int Orthop. 2012 Jun;36(6):1255-60. doi: 10.1007/s00264-011-1470-9. Epub 2012 Jan 22. PMID 22270861
- [Background] Reis T, Schneider F, Welzel G, Schmidt R, Bludau F, Obertacke U, Wenz F. Intraoperative radiotherapy during kyphoplasty for vertebral metastases (Kypho-IORT): first clinical results. Tumori. 2012 Jul-Aug;98(4):434-40. doi: 10.1177/030089161209800406. PMID 23052158
- [Background] Bludau F, Welzel G, Reis T, Schneider F, Sperk E, Neumaier C, Ehmann M, Clausen S, Obertacke U, Wenz F, Giordano FA. Phase I/II trial of combined kyphoplasty and intraoperative radiotherapy in spinal metastases. Spine J. 2018 May;18(5):776-781. doi: 10.1016/j.spinee.2017.09.011. Epub 2017 Sep 28. PMID 28962909
- [Background] Sethi A, Emami B, Small W Jr, Thomas TO. Intraoperative Radiotherapy With INTRABEAM: Technical and Dosimetric Considerations. Front Oncol. 2018 Mar 26;8:74. doi: 10.3389/fonc.2018.00074. eCollection 2018. PMID 29632850
- [Background] Bludau F, Welzel G, Reis T, Abo-Madyan Y, Sperk E, Schneider F, Clausen S, Ruder AM, Obertacke U, Ghaly MM, Wenz F, Giordano FA. Combined kyphoplasty and intraoperative radiotherapy (Kypho-IORT) versus external beam radiotherapy (EBRT) for painful vertebral metastases - a randomized phase III study. BMC Cancer. 2019 May 9;19(1):430. doi: 10.1186/s12885-019-5666-5. PMID 31072314
- [Result] Bludau F, Winter L, Welzel G, Obertacke U, Schneider F, Wenz F, Ruder AM, Giordano FA. Long-term outcome after combined kyphoplasty and intraoperative radiotherapy (Kypho-IORT) for vertebral tumors. Radiat Oncol. 2020 Nov 12;15(1):263. doi: 10.1186/s13014-020-01715-z. PMID 33183307